CLINICAL TRIAL: NCT04654559
Title: Development of a Fever Detection Algorithm Based on Non-invasive Skin-based Sensor Values in Infants up to 18 Months of Age
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Temporary stop & analyze current data. Study may be resumed.
Sponsor: greenTEG AG (Industry)
Collaborators: University Children's Hospital, Zurich (Other); Department of Child Development, Children's Hospital St. Gallen, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6058_Baby_study_1
Record Dates: First submitted 2020-11-26; First posted 2020-12-04 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Fever
Keywords: core body temperature; fever; wearable
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unobtrusive data collection (Other)
  Interventions: Other: Unobtrusive data collection using wearable non-invasive sensors

INTERVENTIONS:
Other: Unobtrusive data collection using wearable non-invasive sensors — Two wearable non-invasive sensors will be mounted to the patients skin (lateral rib cage and foot). These wearable non-invasive sensors are measuring unobtrusively skin based parameters (no diagnosis will be made), which will be used for fever detection algorithm development..

SUMMARY:
Fever of infants up to 18 months of age will be monitored in the hospital using the standard clinical methods and wearable research prototypes. These research prototypes will be measuring continuously and non-invasively skin based parameters, with which the feasibility of developing a fever detection algorithm will be investigated.

DETAILED DESCRIPTION:
Background and Rationale:

In daily clinical practice, core body temperature (CBT) of infants with fever symptoms is monitored using sporadic rectal measurements. Because these sporadic invasive measurements are time consuming for the medical staff and displeasing for patients, an alternative method to assess CBT/fever is needed. The company greenTEG is developing a CBT algorithm which calculates CBT continuously form skin temperature (ST), corresponding heat flux (HF) and other skin-based parameters. The algorithm development will be achieved by collecting skin-based parameters and reference CBT values from infants having fever in a clinical setting.

Objective(s):

Develop and validate an algorithm that allows the detection of fever in infants through a non-invasive sensor system, which calculates CBT from ST, HF and other skin-based data streams, allowing a more effective patient management.

Statistical Considerations:

The measures of quality will be: 1) The mean absolute difference (MAD) between the CBT prediction and the reference signal where the mean is taken over the whole measurement of a single patient. An aggregate performance measure over a group of patients is defined by averaging the MAD values of each patient in the group. 2) the 2σ (standard deviation) range of the Bland-Altmann-Plot between the CBT prediction and the reference signal. This is calculated either for individual patient data or for the combined data of all patients together. As we have defined a group of patients for algorithm validation, the total improvement will be defined by comparing the above aggregate performance measures of old and new algorithm for the validation group. We expect the factors age, sex to influence the algorithmic prediction. Balancing the probability of occurrence of the factors in the population and the overall size of the study, a final size of 50 patients is reasonable.

Study procedures:

Infants will be recruited and screened 1 days before the measurements starts. Two research prototypes will be applied to the patient on the left side of the body (lateral ribcage and foot), after being admitted to the hospital and parents having signed the informed consent. For all infants rectal measurement will be asses every 8 hours, as reference temperature. For infants older than 6 months, in addition to rectal temperature, ear temperature will be assessed every 4 hours with an infrared ear thermometer. The whole measurement procedure will last 18-72 hours, depending on the stationary stay of the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* Infants from two weeks after birth and due date up to 18 months of age
* Infants which are staying at the Nursery and the University Children's Hospital Zurich or Children's Hospital of Eastern Switzerland, St. Gallen for more than 1 day
* Informed consent signed by parents or by legal representatives

Exclusion Criteria:

* Acute medical contradiction against medical plaster and adhesives (e.g. skin diseases or allergies).
* Irritated or damaged skin (e.g. burn, rush, eczema)
* Infant with congenital anomalies (e.g. malformations of the anus)
* Disease or brain injury which cause a disturbance of the thermoregulation
* Comatose infant's
* Infants with implants (e.g. pacemaker, cochlear implants)

Ages: 2 Weeks to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Continuous and non-invasive skin temperature at the lateral rib cage position | Participants will be monitored continuously and unobtrusively with the research prototypes over a 1-3 day time period, depending on the stationary stay in the hospital
  Skin temperature data collected continuously and non-invasively using a research prototype at the lateral ribcage. The skin temperature is measured directly underneath the research prototype on the surface of the skin in degree Celsius.
Continuous and non-invasive heat flux at the lateral rib cage position | Participants will be monitored continuously and unobtrusively with the research prototypes over a 1-3 day time period, depending on the stationary stay in the hospital
  Heat flux data collected continuously and non-invasively using a research prototype at the lateral ribcage. Most of this heat flux will be the thermal energy transmitted from the participants body and is measured in watts per square meters.
Continuous and non-invasive skin temperature at the foot position | Participants will be monitored continuously and unobtrusively with the research prototypes over a 1-3 day time period, depending on the stationary stay in the hospital
  Skin temperature data collected continuously and non-invasively using a research prototype at the foot. The skin temperature is measured directly underneath the research prototype on the surface of the skin in degree Celsius.
Continuous and non-invasive heat flux at the lateral foot position | Participants will be monitored continuously and unobtrusively with the research prototypes over a 1-3 day time period, depending on the stationary stay in the hospital
  Heat flux data collected continuously and non-invasively using a research prototype at the foot. Most of this heat flux will be the thermal energy transmitted from the participants body and is measured in watts per square meters.
Sporadic rectal temperature measurement | Every 8 hours over a 1-3 day time period, depending on the stationary stay in the hospital
  Rectal temperature will be measured every 8 hours by medical staff using the clinically established method of the hospital. This is a standard clinical routine and the precise timing of this measurement is determined by the medical staff according to their daily work routine.
Sporadic ear temperature measurements | Every 4 hours over a 1-3 day time period, depending on the stationary stay in the hospital
  For infants older than 6 months of age only: Ear temperature will be measured every 4 hours using an infrared ear thermometer. The every second ear temperature measurement will coincide with the rectal temperature measurement.

SECONDARY OUTCOMES:
Heart rate | Participants will be monitored continuously and unobtrusively with the research prototypes over a 1-3 day time period, depending on the stationary stay in the hospital
  Heart rate [beats per minute] will be collected using the research prototype on the foot
SpO2 | Participants will be monitored continuously and unobtrusively with the research prototypes over a 1-3 day time period, depending on the stationary stay in the hospital
  Oxygen saturation (SpO2) will be collected using the research prototype on the foot

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Berger, Prof. Dr., Principal Investigator — University Children's Hospital, Zurich
Locations (2):
- Switzerland (2):
  - Children's Hospital of Eastern Switzerland, St. Gallen, Sankt Gallen
  - University Children's Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided
The results of this study will be published in a suited journal. Publication strategy is still in discussion.